CLINICAL TRIAL: NCT02908087
Title: Incretin-based Therapy in Early Diagnosed Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Oulu University Hospital (Other); Tampere University Hospital (Other); Turku University Hospital (Other Government); Skane University Hospital (Other)
Responsible Party: Principal Investigator, Riitta Veijola, Professor, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LiraT1D10-30; 2014-004760-37 (EudraCT Number); 3-SRA-2014-301-M-R (Other Grant/Funding Number: Juvenile Diabetes Research Foundation International); U1111-1177-0661 (Other: WHO)
Record Dates: First submitted 2016-09-06; First posted 2016-09-20 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Type 1 Diabetes
Keywords: Diabetes Type 1; Diabetes, Insulin-Dependent; Liraglutide; GLP-1 Analogue; Early diagnosis
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Disease | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Victoza® (liraglutide) (Active Comparator): Subjects with early diagnosis of type 1 diabetes (no symptoms, diagnosis in OGTT) aged 10-30 years, and treated with insulin are treated with Victoza®
  Interventions: Drug: Victoza® (liraglutide)
- Placebo (Placebo Comparator): Subjects with early diagnosis of type 1 diabetes (no symptoms, diagnosis in OGTT) aged 10-30, and treated with insulin are treated with placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Victoza® (liraglutide) — Daily subcutaneous injections with increasing doses up to 1.8 mg per day. Duration of treatment 6 months. Duration of follow-up 6 months.
  Arms: Victoza® (liraglutide)
Drug: Placebo — Daily subcutaneous injections with increasing doses up to 1.8 mg per day. Duration of treatment 6 months. Duration of follow-up 6 months.
  Arms: Placebo

SUMMARY:
The main objective of the trial is to study whether daily treatment with liraglutide improves insulin secretion and reduces the requirement of exogenous insulin, and whether liraglutide treatment is tolerable and safe in subjects aged 10-30 years, having an early diagnosis of type 1 diabetes (no symptoms, diagnosis in OGTT), and treated with insulin.

ELIGIBILITY:
Inclusion Criteria:

* 10-30 years of age
* early diagnosis type 1 diabetes (no symptoms, diagnosis in OGTT)
* not pregnant.

Exclusion Criteria:

* allergic to liraglutide or other ingredients of Victoza®
* diabetic ketoacidosis
* previous treatment in the last three months with any antidiabetic medication other than insulin
* impaired liver or kidney function or on dialysis
* severe heart failure
* severe stomach or gut problem resulting in gastroparesis, or inflammatory bowel disease
* past or current history of pancreatitis
* serum calcitonin value above normal (>50 ng/l or ≥3.4pmol/l)
* presence of any chronic metabolic, hematologic or malignant disease
* obesity BMI ≥30
* pregnant females and females of childbearing potential who are not using adequate contraceptive methods.
* breast-feeding

Ages: 10 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2016-03; Primary Completion 2021-05 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Serum C-peptide AUC | From baseline to 26 and 52 weeks
  Serum C-peptide area under the curve (AUC) during 2-hour MMTT (mixed-meal tolerance test)

SECONDARY OUTCOMES:
Safety: Serum and urine amylase, serum lipase, serum calcitonin levels will be monitored | From baseline to 26 and 52 weeks
  Safety: Serum and urine amylase, serum lipase, serum calcitonin levels will be monitored during the 26 weeks treatment period and 26 weeks follow-up period
Number of hypoglycemia episodes | From baseline to 26 and 52 weeks
  Number of hypoglycemia episodes during the 26 weeks treatment period and 26 weeks follow-up period
Frequency of gastrointestinal side effects | 12 months
  Frequency of gastrointestinal side effects (diarrhea, nausea, vomiting) during the 26 weeks treatment period and 26 weeks follow-up period
Insulin dose | From baseline to 26 and 52 weeks
  Insulin dose IU/kg/day

CONTACTS AND LOCATIONS:
Overall Officials: Riitta Veijola, MD, Principal Investigator — University of Oulu
Locations (4):
- Finland (3):
  - University of Oulu and Oulu University Hospital, Dept of Children and Adolescents, Oulu
  - University of Tampere and Tampere University Hospital, Tampere
  - University of Turku and Turku University Hospital, Turku
- Lund University and Skåne University Hospital, Malmo, Sweden

REFERENCES:
- [Derived] Kero J, Koskenniemi JJ, Karsikas S, Pokka T, Lou O, Toppari J, Veijola R. INnoVative trial design for testing the Efficacy, Safety and Tolerability of 6-month treatment with incretin-based therapy to prevent type 1 DIAbetes in autoantibody positive participants: A protocol for three parallel double-blind, randomised controlled trials (INVESTDIA). Diabet Med. 2022 Oct;39(10):e14913. doi: 10.1111/dme.14913. Epub 2022 Jul 22. PMID 35797241